CLINICAL TRIAL: NCT06543953
Title: Remote Support for Cochlear Implant Recipients: Evaluation of the HearCare MED-EL App
Acronym: HCARE
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: MED-EL Elektromedizinische Geräte GesmbH (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: MED-EL_CRD_2023_01
Record Dates: First submitted 2024-06-27; First posted 2024-08-09 (Actual); Last update posted 2025-12-01 (Actual); Status verified 2025-11

CONDITIONS: Hearing Loss, Sensorineural; Cochlear Implant
MeSH Terms: conditions — Hearing Loss, Sensorineural

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- HearCare MED-EL App (Other): Subjects perform system check and install audio processor configuration via the HearCare MED-EL App
  Interventions: Device: HearCare MED-EL App

INTERVENTIONS:
Device: HearCare MED-EL App — The main task of the HearCare MED-EL App is to perform technical checks on both implants and audio processors and create backups of audio processor configurations so that these configurations can be written on to an empty audio processor of the same type.

SUMMARY:
This clinical investigation intends to assess safety and performance of the HearCare MED-EL App, a remote care option for recipients of MED-EL cochlear implants

DETAILED DESCRIPTION:
Remote care solutions can provide cochlear implant users a greater convenience, accessibility, and personalized care. These advantages stem from the ability to fine-tune and adjust their devices from the comfort of their own environments, without the need for frequent and time-consuming in-person clinic visits.

Remote care allows clinicians to remotely assess data, provide guidance, and make necessary adjustments, all while minimizing the need for physical presence. This streamlined approach translates to increased capacity for serving a larger number of patients, ultimately leading to improved patient outcomes.

The HearCare MED-EL App is a mobile smartphone application designed for recipients of at least one compatible MED-EL cochlear implant and respective audio processor. The app manages technical checks on compatible cochlear implants and audio processors, creates and utilizes backups of audio processor configurations, and performs updates of audio processor configurations by acting as an executive organ of the MAESTRO System Software. The app reduces face-to-face follow-up appointments of users/caregivers with hearing professionals while maintaining safe and ongoing care for all individuals.

This clinical investigation aims to evaluate the HearCare MED-EL App regarding safety and performance.

ELIGIBILITY:
Inclusion Criteria:

* Age > 18 years
* Implanted with at least one MED-EL Cochlea Implant (CI) for at least 3 months
* Fitted with at least one audio processor compatible with the HearCare MED-EL App (i.e. SONNET 2, SONNET 2 EAS, RONDO 3 or newer)
* Signed and dated Informed Consent Form (ICF) before the start of any study-specific procedure

Exclusion Criteria:

* Lack of compliance with any inclusion criteria
* Implanted with C40X and C40C
* Implanted with an Auditory Brainstem Implant (ABI) or Split electrode array
* Anything that, in the opinion of the Investigator, would place the subject at increased risk or preclude the subject's full compliance with or completion of the study (e.g. psychological disorders, neurologic or motoric comorbidity that could restrict subjects from using the app)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Actual)
Dates: Start 2024-08-20 (Actual); Primary Completion 2025-11-26 (Actual); Study Completion 2025-11-26 (Actual)

PRIMARY OUTCOMES:
Primary Endpoint to assess performance of the HearCare MED-EL App by installing a new audio processor configuration and performing a system check with the HearCare MED-EL App | immediately after the intervention
  The primary endpoint is success rate of the HearCare MED-EL app in percent for both the installation of new audio processor configurations and the detection of technical issues of audio processors or implants.

SECONDARY OUTCOMES:
Speech test in quiet | immediately after the intervention
  Speech test in quiet results (Freiburg Monosyllables at 65 dB SPL)
Speech test in noise | immediately after the intervention
  Speech test in noise results (adaptive SRT50 measured with Oldenburger Satztest (OLSA)) (optional)
Product specific questionnaire (for users) | 2 months after the intervention
  Results of the product-specific user questionnaire (use of the App and satisfaction with the App). This questionnaire has various questions with different answer options (yes/no; amount of use; Likert scale, open text). Results to each question will be analyzed descriptively.
Product specific questionnaire (for professionals) | through study completion, an average of 2 years
  Results of the product-specific professional user questionnaire (satisfaction, performance, safety, and off-label use) by professionals. This questionnaire has various questions with different answer options (yes/no; amount of use; Likert scale, open text). Results to each question will be analyzed descriptively.
Device parameters | immediately after the intervention
  Readout of device parameters stored in the devices internal memory/cloud services (e.g. log files, battery status, audio processor configurations, system check parameters, usage times)
Incidents of device related adverse events | through study completion, an average of 2 years
  The safety profile of the HearCare MED-EL App will be evaluated through the analysis of device-related adverse events and in particular Unanticipated Serious Adverse Device Effect (USADE) assessment.

CONTACTS AND LOCATIONS:
Overall Officials: Andreas Büchner, Prof., Principal Investigator — Medizinsche Hochschule Hannover
Locations (3):
- Germany (3):
  - Katholisches Klinikum Bochum, Bochum
  - Medizinische Hochschule Hannover, Hanover
  - Universitätsklinikum Würzburg, Würzburg